CLINICAL TRIAL: NCT01126424
Title: A Study to Compare the Cognitive Effect of Solifenacin 5mg Once-daily and Oxybutynin 5mg Twice-daily After Chronic Dosing Versus Placebo in Subjects 75 Years and Over With Mild Cognitive Impairment - A Double-blind, Randomized, Multi-center Study
Brief Title: A Study to Compare Two Medications With an Inactive Medication and Look at the Effect on a Person's Mental Ability
Acronym: SENIOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 905-EC-008; 2008-005966-29 (EudraCT Number)
Record Dates: First submitted 2010-04-29; First posted 2010-05-19 (Estimated); Results first posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-09

CONDITIONS: Cognition
Keywords: Anti-muscarinics; Anti-cholinergics; Cognition; Solifenacin
MeSH Terms: interventions — Solifenacin Succinate; oxybutynin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Solifenacin (Experimental): Participants received 21 days of treatment with 5 mg solifenacin, in tablet form once a day.
  Interventions: Drug: Solifenacin
- Oxybutynin (Active Comparator): Participants received 21 days of treatment with 10 mg oxybutynin (1 x 5 mg twice daily) in capsule form.
  Interventions: Drug: Oxybutynin
- Placebo (Placebo Comparator): Participants received 21 days of treatment with placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solifenacin — tablet
  Other Names: YM905
  Arms: Solifenacin
Drug: Oxybutynin — capsule
  Arms: Oxybutynin
Drug: Placebo — tablet
  Arms: Placebo

SUMMARY:
The purpose is to compare solifenacin and oxybutynin with an inactive tablet and assess any potential effects on mental ability.

DETAILED DESCRIPTION:
All subjects will receive each intervention during the course of the study. Subjects will complete a 21-day washout period between treatment periods and following last treatment period.

ELIGIBILITY:
Inclusion Criteria:

* The subject has mild cognitive impairment as determined by mini-mental state examination (MMSE) ≥ grade 24
* The subject conforms to the Stockholm criteria for mild cognitive impairment as assessed by the investigator
* The subject has a body mass index (BMI) between 18.0 to 30.0 kg/m2 inclusive
* The subject is available to complete the study

Exclusion Criteria:

* The subject has moderate or severe cognitive impairment as determined by MMSE criteria at screening, ≤ grade 23
* The subject has depression as determined by Geriatric Depression Scale (GDS) short form ≥ 5 at screening
* The subject has a history of urinary retention, severe gastrointestinal obstruction (including paralytic ileus or intestinal atony or toxic megacolon or severe ulcerative colitis), myasthenia gravis, uncontrolled narrow angle glaucoma or shallow anterior chamber or deemed to be at risk for these conditions
* The subject is undergoing hemodialysis or has severe renal impairment or moderate hepatic impairment and who are on treatment with a potent CYP3A4 inhibitor, e.g. Ketoconazole
* The subject has uncontrolled diabetes mellitus
* The subject has a positive pre-study hepatitis B surface antigen, hepatitis C antibody or HIV result at time of screening
* The subject has a history of drug and / or alcohol abuse at time of screening
* The subject has an average weekly alcohol intake of greater than 21 units (male) or 14 units (female) within ≤ 3 months prior to screening (1 unit is 270cc of beer, 40cc of spirits or 125cc of wine)
* The subject has a history of smoking more than 10 cigarettes (or the equivalent amount of tobacco) per day within ≤ 3 months prior to screening
* The subject has a history of known or suspected hypersensitivity to solifenacin succinate, oxybutynin hydrochloride, other anti-cholinergics or lactose, to any component of the dosage form
* The subject has taken any unstable doses of prescribed medication within ≤ 1 month prior to screening or over-the-counter medicine (including vitamins and herbal remedies) within 48 hours prior to the first study day, which in the opinion of the Investigator, will interfere with the study procedures or compromise safety
* The subject is currently dosing with medication(s) intended to treat overactive bladder symptoms or has history of non-drug treatment intended to treat overactive bladder symptoms within ≤ 3 months prior to screening
* The subject has any clinically significant abnormality following Investigator review of the physical examination
* The subject has any clinically significant abnormality following the Investigator's review of the ECG
* The subject has mobility impairment that precludes the assessment of postural stability
* The subject has any clinically significant abnormal heart rate or blood pressure measurements, at the screening visit (dBP > 90mmHg, sBP > 160mmHg or HR < 40bpm or > 100bpm)
* The subject has any clinically significant abnormality following Investigator's review of the biochemistry & hematology results which, in the opinion of the Investigator, contraindicates their participation
* The subject has donated blood or plasma within ≤ 3 months prior to screening or more than 500ml or 1 unit of blood or plasma within ≤ 6 months prior to screening
* The subject, may find it difficult to adhere to the provisions of treatment and observation specified in the protocol
* The subject has participated in any clinical study within ≤ 3 months prior to screening
* The subject has any clinical condition, diagnosis, symptomatology or ongoing investigation, which, contraindicates their participation
* The subject is an employee of Astellas Pharma, Cognitive Drug Research, and any other third party related to the study site

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe Ltd.
Locations (3):
- United Kingdom (3):
  - Blackpool, Lancashire
  - Manchester, Lancashire
  - Bradford, Yorkshire

REFERENCES:
- [Background] Wright BM. A simple mechanical ataxia-meter. J Physiol. 1971 Oct;218 Suppl:27P-28P. No abstract available. PMID 5130616
- [Derived] Wagg A, Dale M, Tretter R, Stow B, Compion G. Randomised, multicentre, placebo-controlled, double-blind crossover study investigating the effect of solifenacin and oxybutynin in elderly people with mild cognitive impairment: the SENIOR study. Eur Urol. 2013 Jul;64(1):74-81. doi: 10.1016/j.eururo.2013.01.002. Epub 2013 Jan 11. PMID 23332882
- See also: Link to Prescribing Information — http://www.astellas.us/docs/vesicare.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Solifenacin / Oxybutynin / Placebo: Participants received 21 days of each treatment in the following order: 5 mg solifenacin, 10 mg oxybutynin, placebo. There was a 21-day washout period between each treatment period.
- Solifenacin / Placebo / Oxybutynin: Participants received 21 days of each treatment in the following order: 5 mg solifenacin, placebo, 10 mg oxybutynin. There was a 21-day washout period between each treatment period.
- Oxybutynin / Placebo / Solifenacin: Participants received 21 days of each treatment in the following order: 10 mg oxybutynin, placebo, 5 mg solifenacin. There was a 21-day washout period between each treatment period.
- Oxybutynin / Solifenacin / Placebo: Participants received 21 days of each treatment in the following order: 10 mg oxybutynin, 5 mg solifenacin, placebo. There was a 21-day washout period between each treatment period.
- Placebo / Solifenacin / Oxybutynin: Participants received 21 days of each treatment in the following order: placebo, 5 mg solifenacin, 10 mg oxybutynin. There was a 21-day washout period between each treatment period.
- Placebo / Oxybutynin / Solifenacin: Participants received 21 days of each treatment in the following order: placebo, 10 mg oxybutynin, 5 mg solifenacin. There was a 21-day washout period between each treatment period.
Period: Overall Study
Arm/Group | Solifenacin / Oxybutynin / Placebo | Solifenacin / Placebo / Oxybutynin | Oxybutynin / Placebo / Solifenacin | Oxybutynin / Solifenacin / Placebo | Placebo / Solifenacin / Oxybutynin | Placebo / Oxybutynin / Solifenacin
Started | 3 (All randomized patients who took at least 1 dose of study drug) | 4 (All randomized patients who took at least 1 dose of study drug) | 5 (All randomized patients who took at least 1 dose of study drug) | 6 (All randomized patients who took at least 1 dose of study drug) | 4 (All randomized patients who took at least 1 dose of study drug) | 4 (All randomized patients who took at least 1 dose of study drug)
Safety Analysis Subset 1 (SAF 1) | 3 (Took at least 1 dose of study drug and completed cognitive function tests for at least 2 treatments.) | 4 (Took at least 1 dose of study drug and completed cognitive function tests for at least 2 treatments.) | 4 (Took at least 1 dose of study drug and completed cognitive function tests for at least 2 treatments.) | 4 (Took at least 1 dose of study drug and completed cognitive function tests for at least 2 treatments.) | 4 (Took at least 1 dose of study drug and completed cognitive function tests for at least 2 treatments.) | 4 (Took at least 1 dose of study drug and completed cognitive function tests for at least 2 treatments.)
Completed | 3 | 4 | 4 | 3 | 2 | 4
Not Completed | 0 | 0 | 1 | 3 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solifenacin / Oxybutynin / Placebo | Solifenacin / Placebo / Oxybutynin | Oxybutynin / Placebo / Solifenacin | Oxybutynin / Solifenacin / Placebo | Placebo / Solifenacin / Oxybutynin | Placebo / Oxybutynin / Solifenacin | Total
Number analyzed (Participants) | 3 | 4 | 5 | 6 | 4 | 4 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 79.7 (3.8) | 78.8 (2.5) | 80.2 (4.4) | 76.7 (2.0) | 79.3 (2.9) | 79.0 (4.1) | 78.8 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 3 | 2 | 2 | 12
  Male | 2 | 3 | 2 | 3 | 2 | 2 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3 | 4 | 5 | 6 | 4 | 4 | 26
Stockholm criteria for mild cognitive impairment [Number; unit: participants] — The Stockholm criteria for identification of mild cognitive impairment are:
  * Cognitive complaints from patients or families
  * Reporting of decline in cognitive functioning relative to previous abilities during the past year by patient or informant
  * Cognitive disorders as evidenced by clinical evaluation (impairment in memory or in another cognitive domain)
  * Absence of major repercussions on daily life (the patient may report difficulties in day-to-day activities)
  * Absence of dementia
  participants
    Yes | 3 | 4 | 5 | 6 | 4 | 4 | 26
    No | 0 | 0 | 0 | 0 | 0 | 0 | 0
Total Mini-Mental State Examination (MMSE) Score [Mean (Standard Deviation); unit: scores on a scale] — The mini-mental state examination (MMSE) provides measures of orientation, registration (immediate memory), short-term memory (but not long-term memory) and language functioning. The investigator reads a series of questions aloud clearly and slowly to the patient and scores each incorrect answer with "0" and each correct answer with "1", for a maximum score of 30.
  scores on a scale | 27.7 (0.58) | 28.3 (1.26) | 28.0 (1.00) | 27.3 (1.75) | 26.5 (1.00) | 27.3 (2.06) | 27.5 (1.39)
Total Geriatric Depression Scale (GDS) Score [Mean (Standard Deviation); unit: scores on a scale] — The short-form geriatric depression scale (GDS) was developed as a basic screening measure for depression in older adults. It is a 15-point questionnaire in which the patient is required to answer 'yes' or 'no'. The GDS responses were translated into a binary scale on which "1" was indicative of depression and "0" was not; the total score ranges from 0 to 15. A score of > 5 points is considered suggestive of depression. Scores of > 10 points are almost always indicative of depression.
  scores on a scale | 1.0 (1.73) | 1.0 (0.82) | 1.4 (1.67) | 1.0 (0.63) | 1.3 (0.96) | 1.8 (1.26) | 1.2 (1.11)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cognitive Function Composite Score - Power of Attention
Description: Cognitive effects were assessed at the end of each treatment period using a computerized assessment system at time points close to the predicted time to attain maximum plasma concentration (Tmax) for solifenacin (6 hours) and oxybutynin (2 hours). Power of attention is calculated from the sum of three cognitive function speed tests: Simple Reaction Time, Choice Reaction Time and the Speed of Detections in Digit Vigilance task. A low score reflects a fast reaction time and a high intensity of concentration. A positive change from baseline reflects impairment compared to the baseline assessment.
Time Frame: Assessed at each treatment period baseline visit (the day prior to the first dose of each treatment; Days -1, 42, 84) and at the end of each treatment period (Days 21, 63 and 105). At each visit, tests were performed at 2 and 6 hours post-dose.
Population: The number of participants analyzed represents the Safety Analysis Subset 1 (SAF1), consisting of all randomized patients who took at least one dose of the study medication and who completed the cognitive function tests for at least two treatment periods. The number of participants per arm is consistent for all categories / rows of the data table.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Solifenacin | Oxybutynin | Placebo
Number analyzed (Participants) | 22 | 20 | 22
msec
  Baseline at 2 hours [Oxybutynin Tmax] | 1413.67 (180.242) | 1423.38 (186.163) | 1401.21 (177.194)
  Change from Baseline at 2 hours | -5.86 (71.371) | 17.81 (92.340) | 1.99 (54.145)
  Baseline at 6 hours [Solifenacin Tmax] | 1421.80 (191.303) | 1405.41 (182.929) | 1393.98 (189.128)
  Change from Baseline at 6 hours | -14.80 (87.918) | -0.74 (62.650) | 11.77 (93.655)
Statistical Analysis 1: Comparison: Solifenacin vs Placebo; Comparison of solifenacin versus placebo change from Baseline at 6 hours The null hypothesis was that the mean change from baseline was the same in both treatments; Test type: Superiority or Other; p = 0.3771, ANCOVA; The analysis was performed using an ANCOVA model with fixed effect for treatment, period, subjects as a random effect and baseline as a covariate; Least Square Mean Difference = -20.986, 95% CI 2-sided [-68.580 to 26.607]
Statistical Analysis 2: Comparison: Oxybutynin vs Placebo; Comparison of oxybutynin versus placebo change from Baseline at 2 hours The null hypothesis was that the mean change from baseline was the same in both treatments; Test type: Superiority or Other; p = 0.4487, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = 17.508, 95% CI 2-sided [-28.854 to 63.870]

2. Secondary Outcome: Change From Baseline in Postural Stability Test
Description: The postural stability test measures the ability to stand upright without moving, and was assessed at the end of each treatment period using a computerized assessment system at time points close to the predicted time to attain maximum plasma concentration for solifenacin and oxybutynin. Using apparatus modeled on the Wright Ataxia-meter, a cord from the meter is attached to the patient who is required to stand as still as possible with feet apart and eyes closed for 1 minute.
  The amount of sway is expressed as the total angular movement, summed regardless of sign, in the antero-posterior plane and calibrated in units of one-third degree of angle of sway. Wright (1971) described a range of 20-30 units as a normal range for adults with eyes wide open, increasing by 50 to 100% with eyes shut.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/3 degree of angle of sway
Arm/Group | Solifenacin | Oxybutynin | Placebo
Number analyzed (Participants) | 22 | 20 | 22
1/3 degree of angle of sway
  Baseline at 2 hours [Oxybutynin Tmax] | 37.7 (23.35) | 36.2 (20.05) | 37.5 (20.04)
  Change from Baseline at 2 hours | 5.2 (9.65) | 2.7 (17.04) | 0.4 (16.81)
  Baseline at 6 hours [Solifenacin Tmax] | 37.7 (19.42) | 38.9 (23.59) | 40.0 (26.19)
  Change from Baseline at 6 hours | 9.9 (16.14) | 0.7 (17.60) | -0.1 (10.64)
Statistical Analysis 1: Comparison: Solifenacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0505, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = 9.152, 95% CI 2-sided [-0.023 to 18.326]
Statistical Analysis 2: Comparison: Oxybutynin vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6753, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = 1.846, 95% CI 2-sided [-7.020 to 10.713]

3. Primary Outcome: Change From Baseline in Cognitive Function Composite Score - Continuity of Attention
Description: Cognitive effects were assessed using a computerized assessment system at time points close to the predicted time of maximum plasma concentration for solifenacin and oxybutynin. For continuity of attention, the number of correct responses (out of 50) for choice reaction time was added to the total number of targets correctly identified (out of 45) digit vigilance minus the number of false alarms (total score of -45 to 95). A high score reflects someone able to keep his/her mind on a single task for a prolonged period. A negative change from baseline reflects impairment compared to baseline.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Solifenacin | Oxybutynin | Placebo
Number analyzed (Participants) | 22 | 20 | 22
Scores on a scale
  Baseline at 2 hours [Oxybutynin Tmax] | 91.591 (3.2462) | 91.300 (2.5775) | 91.364 (2.3409)
  Change from Baseline at 2 hours | 0.545 (2.0637) | 0.150 (3.2653) | 0.909 (2.6168)
  Baseline at 6 hours [Solifenacin Tmax] | 91.228 (2.0454) | 91.901 (2.4040) | 91.728 (3.6929)
  Change from Baseline at 6 hours | -0.318 (2.7143) | 0.100 (2.7121) | -0.045 (3.4566)
Statistical Analysis 1: Comparison: Solifenacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5684, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -0.507, 95% CI 2-sided [-2.293 to 1.279]
Statistical Analysis 2: Comparison: Oxybutynin vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2348, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -0.792, 95% CI 2-sided [-2.122 to 0.538]

4. Primary Outcome: Change From Baseline in Cognitive Function Composite Score - Quality of Working Memory
Description: Cognitive effects were assessed at the end of each treatment period using a computerized assessment system at time points close to the predicted time to attain maximum plasma concentration (Tmax) for solifenacin (6 hours) and oxybutynin (2 hours). Quality of working memory is calculated from the sum of two cognitive function sensitivity tests: Numeric Working Memory Sensitivity and Spatial Working Memory Sensitivity, and ranges from -2 to 2. A higher score reflects a good working memory and a negative change from baseline reflects impairment compared to the baseline assessment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Solifenacin | Oxybutynin | Placebo
Number analyzed (Participants) | 22 | 20 | 22
Scores on a scale
  Baseline at 2 hours [Oxybutynin Tmax] | 1.7921 (0.24313) | 1.7251 (0.31582) | 1.7087 (0.24215)
  Change from Baseline at 2 hours | -0.0867 (0.39254) | -0.0043 (0.35428) | 0.0492 (0.37776)
  Baseline at 6 hours [Solifenacin Tmax] | 1.6666 (0.35805) | 1.6441 (0.34113) | 1.7548 (0.35808)
  Change from Baseline at 6 hours | 0.0580 (0.46462) | 0.0633 (0.46684) | 0.0047 (0.41656)
Statistical Analysis 1: Comparison: Solifenacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6275, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -0.040, 95% CI 2-sided [-0.208 to 0.127]
Statistical Analysis 2: Comparison: Oxybutynin vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5361, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -0.046, 95% CI 2-sided [-0.194 to 0.103]

5. Primary Outcome: Change From Baseline in Cognitive Function Composite Score - Quality of Episodic Secondary Memory
Description: Cognitive effects were assessed at the end of each treatment period using a computerized assessment system at time points close to the predicted time of maximum plasma concentration for solifenacin and oxybutynin. Quality of episodic secondary memory is calculated from the sum of 4 tests: Immediate and delayed word recall, and word and picture recognition, and ranges from -200 to 400. A high score reflects a good ability to store, hold and retrieve information of an episodic nature (i.e. an event or a name) and a negative change from baseline reflects impairment compared to baseline.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Solifenacin | Oxybutynin | Placebo
Number analyzed (Participants) | 22 | 20 | 22
Scores on a scale
  Baseline at 2 hours [Oxybutynin Tmax] | 111.893636 (48.525110) | 107.666333 (55.168759) | 110.000152 (51.736947)
  Change from Baseline at 2 hours | -3.788636 (35.609118) | -0.917833 (28.198821) | 0.531515 (42.576179)
  Baseline at 6 hours [Solifenacin Tmax] | 101.363485 (44.919411) | 104.917167 (50.380503) | 106.515000 (45.147568)
  Change from Baseline at 6 hours | 7.728182 (30.836915) | -3.502000 (48.822365) | 1.589394 (35.687431)
Statistical Analysis 1: Comparison: Solifenacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6315, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = 4.655, 95% CI 2-sided [-14.858 to 24.167]
Statistical Analysis 2: Comparison: Oxybutynin vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8670, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -1.457, 95% CI 2-sided [-18.976 to 16.062]

6. Primary Outcome: Change From Baseline in Cognitive Function Composite Score - Speed of Memory
Description: Cognitive effects were assessed at the end of each treatment period using a computerized assessment system at time points close to the predicted time to attain maximum plasma concentration for solifenacin and oxybutynin. Speed of Memory was calculated from the sum of 4 cognitive function speed tests: numeric and spatial working memory and word and picture recognition. A low score reflects that a person is able to recall a name, a face or any other item fast from the episodic secondary memory; a positive change from baseline reflects impairment compared to baseline.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Solifenacin | Oxybutynin | Placebo
Number analyzed (Participants) | 22 | 20 | 22
msec
  Baseline at 2 hours [Oxybutynin Tmax] | 4505.96 (957.434) | 4545.75 (789.173) | 4741.30 (820.101)
  Change from Baseline at 2 hours | 24.09 (762.881) | -11.56 (571.131) | -240.62 (471.516)
  Baseline at 6 hours [Solifenacin Tmax] | 4496.65 (653.186) | 4606.51 (846.669) | 4655.29 (923.390)
  Change from Baseline at 6 hours | -149.79 (494.835) | -118.14 (471.318) | -126.04 (728.870)
Statistical Analysis 1: Comparison: Solifenacin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5953, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -77.919, 95% CI 2-sided [-372.814 to 216.976]
Statistical Analysis 2: Comparison: Oxybutynin vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3526, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = 157.783, 95% CI 2-sided [-182.015 to 497.581]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected by treatment period from first administration of the study/comparative drug until within 7 days of taking the last dose.
Description: A treatment period consists of about 21 treatment days with a follow-up of either about 21 washout days prior to start of next treatment period or a follow-up of 7 days for the last treatment period.
Arm/Group | Solifenacin | Oxybutynin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/25 | 0/22
Other Adverse Events (participants affected / at risk) | 5/23 | 14/25 | 6/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Solifenacin (N=23) | Oxybutynin (N=25) | Placebo (N=22)
Vitreous detachment (Eye disorders) | 1 | 0 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Solifenacin (N=23) | Oxybutynin (N=25) | Placebo (N=22)
Dry mouth (Gastrointestinal disorders) | 4 | 13 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Balance disorder (Nervous system disorders) | 2 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may not publish trial data generated at their specific study site without prior written approval of the Sponsor.